CLINICAL TRIAL: NCT03849573
Title: A Mindfulness-Based e-Health Intervention to Improve Medication Adherence Among Breast Cancer Survivors
Brief Title: A Web-Based Tool to Improve Breast Cancer Survivorship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Betina Yanez, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00206180
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Hormone Dependent Neoplasms; Adherence to Hormone Therapy
Keywords: eHealth; Adherence; Health Related Quality of Life; Symptom Burden; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Hormone-Dependent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction + Hormone Therapy Education (Experimental)
  Interventions: Behavioral: "OncoTool" Intervention (MBSR + HT education)
- Hormone Therapy Education + Overall Health Education (Active Comparator)
  Interventions: Behavioral: "Oncotool" Control (health +HT education)

INTERVENTIONS:
Behavioral: "OncoTool" Intervention (MBSR + HT education) — OncoTool is a website intended to improve self-management practices for helping cancer patients cope with stress and improve health-related quality of life. OncoTool provides mindfulness-based education and management for dealing with the numerous physical and mental side effects associated with hormone therapy (e.g., muscle and joint pain, vaginal dryness, depressive symptoms). OncoTool is a website designed to improve hormone therapy adherence by improving quality of life, and hormone therapy associated symptom burden. Both intervention and active comparator conditions are administered to participants for 8 weeks.
  Arms: Mindfulness-based stress reduction + Hormone Therapy Education
Behavioral: "Oncotool" Control (health +HT education) — OncoTool is a health promotion website with health education on subjects like nutrition and exercise specific to breast cancer survivors, as well as general advice on lifestyle choices and prevention. The Oncotool control has similar HT education content as the experimental content but without the CBT and MBSR state. Both intervention and active comparator conditions are administered to participants for 8 weeks.
  Arms: Hormone Therapy Education + Overall Health Education

SUMMARY:
The purpose of this study is to examine the efficacy of a psychosocial eHealth intervention on the proposed primary outcomes, hormone therapy adherence and health related quality of life (HRQoL), in breast cancer survivors.

The intervention components include mindfulness-based stress reduction, breast cancer knowledge, stress awareness and management, social support, and enhanced communication. The intervention will be delivered via an online application over an 8-week period.

Participants are randomized into either an intervention application (described above) or a control application (health information and general health promotion strategies). Aside from having access to the online application for the recommended 8 weeks with weekly online focus groups, participation in this study includes four assessments: baseline (at the beginning of the research study), post-intervention (8 weeks after baseline), a 6-month follow-up and a 12-month follow-up.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer among women in the U.S. Approximately 75% to 80% of breast cancer survivors are prescribed HT (hormone therapy) medication for 5 to 10 years following primary treatment. Five years of adjuvant HT among women with non-metastatic cancer reduces the risk of recurrences by 50%. Adherence to HT is also an independent predictor of breast cancer mortality, reducing the risk by up to 28%. HT-side effects, however, are not only a major source of distress but also among the most robust predictors of non-adherence to HT. Therefore, effective management and ability to reduce the burden of these side effects are critically important to achieve optimal HT adherence. Because HT side effects may persist for years and are not easily managed, MBSR's mind-body approach and emphasis on non-judgmental attitudes, acceptance, and uncertainty tolerance may be an especially beneficial approach to helping cancer survivors cope with the burdensome medication-related side effects, thus improving adherence to medication. The investigators propose that a mindfulness-based stress reduction (MBSR) intervention that has been efficacious in reducing HT side effects and improving HRQoL in cancer patients may also prove beneficial in improving HT adherence. After developing a web-based MBSR intervention and refining it via a usability trial, this study will establish the feasibility of a web-delivered, group based MBSR intervention to improve HT medication adherence and HRQoL in patients being treated for breast cancer. It is hypothesized that participants assigned to the MBSR intervention will have better primary outcomes than participants in the control group, which receives standard health information.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. English-speaking (6th grade reading level) as required to complete assessments
3. medical chart confirmed diagnosis of hormone-receptor positive non-metastatic breast cancer
4. Stages I-IIIa
5. completion of any combination of surgical, radiation, and chemotherapy treatment
6. willingness to be randomized into study
7. have initiated HT within the past 6 months as data in literature indicates that the overwhelming majority of women who initiated HT are still adherent within the first 4 months
8. first-time diagnosis of breast cancer
9. access to a computer or tablet with Internet capabilities

Exclusion Criteria:

1. Visual, hearing, voice, or motor impairment that would prevent completion of study procedures
2. diagnosis of an unmanaged psychotic or psychiatric disorder (e.g., clinical depression, anxiety, or PTSD), bipolar disorder, dissociative disorder, or other diagnosis for which participation in this trial is either inappropriate or dangerous - this includes patients who have life-threatening illness (e.g., end-stage kidney disease) or diagnosis of a chronic disease that is associated with a major functional impairment (e.g., chronic severe pain, fibromyalgia)
3. Alzheimer's, dementia or history of stroke

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Self Reported Adherence to Hormone Therapy will be evaluated with the ARMS questionnaire. | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The ARMS (Adherence to Refills and Medications Scale) survey is a previously validated patient-report measure of barriers to medication adherence and adherence-related behavior.
Change in Health Related Quality of Life will be evaluated with The Functional Assessment of Cancer Therapy-Endocrine (FACT-ES) | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The FACT-ES has been used extensively to measure HRQoL. It assesses participant's wellbeing in physical, emotional, social, functional, and concerns specific to endocrine therapy in the last seven days using a five-point response scale.
Electronically Verified Hormone Therapy Adherence will be measured using medication event monitoring systems (MEMS) | MEMS data will be collected continuously during study participation from T1 (prior to starting intervention) to T4 (12 months post-intervention)
  A MEMS cap is an electronic bottle cap that tracks when participants open their medication bottle. MEMS cap data will be collected continuously during the duration of participation in the study.
Pharmacy reported Adherence to Hormone Therapy will be measured using pharmacological records | T4 (12 months post intervention)
  Pharmacy data will be pulled once at approximately T4 when a participant finishes the study. This data will inform how frequently patients refill their hormone therapy medication.

SECONDARY OUTCOMES:
Cancer-Specific Distress will be evaluated using The Impact of Event Scale (IES) | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The IES is made up of two subscales measuring the frequency of intrusion and avoidance experiences after a stressful event. The IES has been widely used among patients diagnosed with cancer.
Breast Cancer Related Knowledge will be evaluated with the Knowledge about Breast Cancer Questionnaire | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  This questionnaire has been tested and validated with breast cancer patients. It is made up of 16 true and false questions regarding general breast cancer knowledge.
Breast Cancer Related Communication and Attitudinal Self Efficacy will be evaluated using the Communication and Attitudinal Self-Efficacy scale for cancer (CASE-cancer) | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The CASE-cancer questionnaire is made up various subscales measuring breast cancer related communication and attitudinal self-efficacy. Each question asks participants to use a four-point response scale to agree or disagree with statements regarding their level of confidence with different skills.
Stress Management Skills will be evaluated with the Brief COPE Inventory | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The Brief COPE is made up of various subscales measuring different ways of coping. Each question as participants to rate how often they have used each coping mechanism in response to their breast cancer experience.
Perceived benefits and cost barriers to using hormone therapy will be assessed using a Beliefs about Medicines scale | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The 11 point Beliefs about Medicines questionnaire assesses patients' beliefs about the efficacy of their treatment as well as their beliefs about how the benefits and side affects of hormone therapy affect their life.
Self-Reported Negative Mood is measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression questionnaire | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The PROMIS Depression questionnaire is a computer adaptive assessment that measures patients' self-reported level of negative mood within the past 7 days.
Emotional Social Support is assessed using the emotional subscale portion of the Medical Outcomes Study - Social Support Survey Instrument (MOS-SSS) | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The 8 question MOS-SSS scale was developed by RAND Healthcare to assess the degree of companionship, assistance, or other types of social support that participants have access to. This study will use the 8 question emotional-informational support subsection.
Patient Self-Efficacy in managing side effects is measured using the PROMIS Self Efficacy for Managing Symptoms | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The PROMIS Self Efficacy for Managing Symptoms survey is a validated, computer adaptive survey to assess how confident participants are in their ability to manage their symptoms and side effects
Mindfulness will be assessed using questionnaires tailored to MBSR treatment | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The Intolerance of Uncertainty, Rumination and Reassure Me survey assesses participants' development in MBSR intervention targets, which will help isolate and assess the effect of MBSR treatment
Concerns about cancer recurrence will be measured using the Concerns about Recurrence scale | T1 (prior to starting intervention), T2 (8 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post intervention)
  The Concerns about Recurrence scale is a 4 question scale that assesses the frequency and intensity of patients' concerns about cancer recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Betina Yanez, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with any researchers outside Northwestern.

DOCUMENTS (1):
  • Informed Consent Form (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT03849573/ICF_000.pdf